CLINICAL TRIAL: NCT02563171
Title: Effects of Non-Surgical Periodontal Treatment on the Gingival Crevicular Fluid Levels of Vaspin and Omentin-1 in Obese Patients With Chronic Periodontitis
Brief Title: Gingival Crevicular Fluid Vaspin and Omentin Levels in Obese Patients With Chronic Periodontitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Umut BALLI (Other)
Responsible Party: Sponsor-Investigator, Umut BALLI, Bulent Ecevit University, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-115-17/06
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Obesity; Periodontitis
Keywords: visceral adipose-specific serpin; intelectin 1 (omentin); Tumor Necrosis Factor-alpha
MeSH Terms: conditions — Obesity; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy periodontium without obesity (Placebo Comparator): GCF samples were taken at baseline Intervention: Gingival crevicular fluid collection
  Interventions: Other: Gingival crevicular fluid collection
- Chronic periodontitis without obesity (Active Comparator): GCF samples were taken before and after treatment chronic periodontitis patients.
  Intervention: Non- surgical periodontal treatment (SRP and oral hygiene instructions)
  Interventions: Other: non surgical periodontal treatment
- Healthy periodontium with obesity (Placebo Comparator): GCF samples were taken at baseline Intervention: Gingival crevicular fluid collection
  Interventions: Other: Gingival crevicular fluid collection
- Chronic periodontitis with obesity (Active Comparator): GCF samples were taken before and after treatment chronic periodontitis patients.
  Intervention: Non- surgical periodontal treatment (SRP and oral hygiene instructions)
  Interventions: Other: non surgical periodontal treatment

INTERVENTIONS:
Other: non surgical periodontal treatment — 1. SRP under local anaesthesia, in a total of 2-3 clinical visits.
  2. Oral hygiene instructions including the modified Bass technique, regular toothpaste, and an appropriate interdental cleaning device with dental floss and interdental brush.
  Arms: Chronic periodontitis with obesity; Chronic periodontitis without obesity
Other: Gingival crevicular fluid collection — GCF collection with filter paper (Periopaper) using the intracrevicular method.
  Arms: Healthy periodontium with obesity; Healthy periodontium without obesity

SUMMARY:
Our objective in this case-control intervention study, therefore, was to explore the effect of nonsurgical periodontal therapy on the GCF levels of vaspin and omentin in patients with chronic periodontitis in order to determine the usefulness of vaspin and omentin as a diagnostic and prognostic biomarker of periodontal disease.

DETAILED DESCRIPTION:
All individuals underwent a full-mouth periodontal examination, which included probing pocket depth (PPD), clinical attachment level (CAL), plaque index (PI), gingival index (GI), bleeding on probing (BOP). BMI and WHR were used for assessing obesity. In addition, HbA1c and fasting plasma glucose levels were used for elimination of diabetes mellitus. Based on the periodontal and anthropometric measurements, individuals (n=76) were divided into four groups: the periodontal-healthy group (n=19), chronic periodontitis group (n=19), periodontal-healthy with obesity group (n=19) and chronic periodontitis with obesity group (n=19). Periodontitis patients received nonsurgical periodontal therapy. GCF sampling and clinical periodontal parameters were assessed before and 6 weeks after therapy. Vaspin, omentin, and TNF-α levels were measured by enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

1-) 30-49 years of age 2-) had a minimum of 20 natural teeth, excluding third molars 3) glycosylated hemoglobi levels <6% 4) fasting plasma glucose levels <100 mg/dl. 5-) Criteria for the periodontal healthy group were GI = 0, PPD≤ 3 mm, and no signs of attachment and bone loss by clinical and radiographic examination.

6-) Criteria for the chronic periodontitis group were clinical signs of inflammation (red color and swelling of the gingival margin), GI ≥ 2, PPD and CAL ≥ 5 mm, and bone loss affecting >30% of the existing teeth on clinical and radiographic examination.

7-) Criteria for obese groups were 30≤ BMI <40 kg/m2, and concomitant WHR ≥0.85 for females and WHR ≥0.90 for males.

8-) Criteria for normal-weight groups were 20≤ BMI <25 kg/m2, and WHR below that determined for obesity.

Exclusion Criteria:

1. Aggressive periodontitis,
2. Periapical pathologies
3. Excessive forces including mechanical forces from orthodontics and occlusion
4. Systemic diseases (e.g., diabetes mellitus; cancer; human immunodeficiency virus; or disorders that could affect adipokines levels and the periodontal conditions)
5. Chronic high-dose steroid therapy, radiation or immunosuppressive therapy
6. Pregnancy, lactation,
7. Smoking within the past five years, or allergy or sensitivity to any drug.
8. Had no history of periodontal therapy or drug therapy (e.g., anti-inflammatories, antibiotics, or any other pharmacological treatment) for at least six months.

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Biochemical parameters (Vaspin and omentin) | Baseline and 6 weeks after treatment
  The changes in levels of vaspin and omentin 6 weeks after periodontal treatment determined by ELISA. The changes in levels of vaspin and omentin were analyzed to determine diagnostic and prognostic potential as a biomarker of periodontal disease.

SECONDARY OUTCOMES:
Tumor necrosis factor alfa | Baseline and 6 weeks after treatment
  The changes in levels of tumor necrosis factor alfa 6 weeks after periodontal treatment determined by ELISA.
Probing pocket depth | Baseline and 6 weeks after treatment
  The changes in probing pocket depth after periodontal treatment.Probing pocket depth was measured for determining severity of disease and clinic outcome.
Clinical attachment level | Baseline and 6 weeks after treatment
  The changes in clinical attachment level after periodontal treatment. Clinical attachment level was measured for determining severity of disease and clinic outcome.
Gingival index | Baseline and 6 weeks after treatment
  The changes in gingival index after periodontal treatment. Gingival index was recorded for classifying and evaluating (coronally) gingival inflammation. Also, gingival index was also analyzed to detect the relationship between vaspin, omentin and tumor necrosis factor alfa.
Plaque index | Baseline and 6 weeks after treatment
  The changes in plaque index after periodontal treatment. Plaque index was recorded for determining and classifying oral hygiene status.
Bleeding on probing | Baseline and 6 weeks after treatment
  The changes in bleeding on probing after periodontal treatment. Bleeding on probing was recorded for classifying and evaluating (apically) gingival inflammation.